CLINICAL TRIAL: NCT03743363
Title: Effects of Exergaming Session Frequency on Work Performance, Cognition, and Mobility in Adults Age 55 to 65
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Principal Investigator, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IKEB009/2018
Record Dates: First submitted 2018-11-06; First posted 2018-11-16 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: balance; movement; exergaming; work performance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergame 3/week (Experimental): The group does active training for 8 weeks after not training.
  Interventions: Other: Exergaming 3/week
- Exergame 2/week (Experimental): The group does active training for 8 weeks after not training.
  Interventions: Other: Exergame 2/week
- Healthy control / Exergame 1/week (Experimental): In the first 8 week-long only control group, The group will do 1 training/week for the next 8 weeks.
  Interventions: Other: Healthy control / Exergaming 1/week

INTERVENTIONS:
Other: Exergame 2/week — virtual training 2 times a week(8 week-long)
  Arms: Exergame 2/week
Other: Exergaming 3/week — virtual training 3 times a week(8 week-long)
  Arms: Exergame 3/week
Other: Healthy control / Exergaming 1/week — In the first 8 week-long only control group. For the next 8 weeks, the control group will do 1 workout per week.
  Arms: Healthy control / Exergame 1/week

SUMMARY:
Aim - determine the immediate and lasting effects of Exergaming frequency on work performance, health, motor, and cognitive function in clerical employees.

DETAILED DESCRIPTION:
Hypothesis - In sedentary clerical workers the introduction of even 1 session / week exercise can cause lasting and correlated improvements in work, motor, and cognitive function, and effect which plateaus at 2 compared with 3 sessions / week. However, 6 months follow up would show residual effects only at the 3/week frequency in those who had become sedentary again.

ELIGIBILITY:
Inclusion Criteria:

* age
* active worker
* no detected neurological status

Exclusion Criteria:

* Sever heart problem
* Sever demeanor
* Alkoholism
* Drug problems

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Motor function | 8 weeks
  Step test (as described by Prieske et al, motion and endurance test)
Motor Function | 8 weeks
  Grip strength - Chair rise (as part of SPPB) the higher score better performance
MOBILITY | 8 weeks
  -SPPB - the higher score better performance
BALANCE Functional reach | 8 weeks
  Beam walking (4, 8, 12 cm 3 trials each, summed distance score) The longer the journey is, the better the performance
Cognitive function | 8 weeks
  - MMSE (questionnaire…) the higher score better performance
Cognitive function | 8 weeks
  - Processing speed: The Digit Symbol Substitution Test (DSST)
Mobility | 8 weeks
  6MWT - The longer the journey is, the better the performance
Mobility | 8 weeks
  Fast gait speed over 10 m - speed, the faster the better
Cognitive function | 8 weeks
  Verbal and visual memory span and working memory (0-100 visual analog sclae-the higher score better performance)

CONTACTS AND LOCATIONS:
Locations (1):
- Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hortobagyi T, Deak D, Farkas D, Blenyesi E, Torok K, Granacher U, Tollar J. Effects of Exercise Dose and Detraining Duration on Mobility at Late Midlife: A Randomized Clinical Trial. Gerontology. 2021;67(4):403-414. doi: 10.1159/000513505. Epub 2021 Mar 3. PMID 33657562